CLINICAL TRIAL: NCT04446663
Title: Toripalimab Combined With Chemoradiotherapy in Locoregionally-advanced Nasopharyngeal Carcinoma: an Open-label, Parallel Controlled, Phase IIa Study
Brief Title: Toripalimab Combined With Chemoradiotherapy in Patients With Locoregionally-advanced Nasopharyngeal Carcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: First People's Hospital of Foshan (Other)
Responsible Party: Principal Investigator, Guo-Yi Zhang, Chief Physician, First People's Hospital of Foshan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JS001-ISS-CO185
Record Dates: First submitted 2020-06-19; First posted 2020-06-25 (Actual); Last update posted 2020-06-25 (Actual); Status verified 2020-06

CONDITIONS: Nasopharyngeal Neoplasms
MeSH Terms: conditions — Nasopharyngeal Neoplasms | interventions — toripalimab; Albumin-Bound Paclitaxel; Cisplatin; Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Toripalimab+induction chemotherapy +CCRT (Experimental): Patients will receive induction chemotherapy with Albumin-bound paclitaxel (260 mg/m2, d1 of every cycle) and cisplatin (80mg/m2, d1 of every cycle), every 3 weeks for 3 cycles before radiotherapy.
  Then patients will receive definitive intensity-modulated radiotherapy (IMRT) of ≥66 Gy（2-2.2Gy/fx）.Concurrent cisplatin of 100mg/m2 will be administered every 3 weeks for 2 cycles during IMRT .
  Toripalimab 240mg will be given every 3 weeks for 6 cycles, started on day 1 of induction chemotherapy
  Interventions: Drug: Toripalimab; Drug: Albumin-bound Paclitaxel; Drug: Cisplatin; Radiation: intensity-modulated radiotherapy
- induction chemotherapy +CCRT (Active Comparator): Patients will receive induction chemotherapy with Albumin-bound paclitaxel (260 mg/m2, d1 of every cycle) and cisplatin (80mg/m2, d1 of every cycle), every 3 weeks for 3 cycles before radiotherapy.
  Then patients will receive definitive intensity-modulated radiotherapy (IMRT) of ≥66 Gy（2-2.2Gy/fx）.Concurrent cisplatin of 100mg/m2 will be administered every 3 weeks for 2 cycles during IMRT .
  Interventions: Drug: Albumin-bound Paclitaxel; Drug: Cisplatin; Radiation: intensity-modulated radiotherapy

INTERVENTIONS:
Drug: Toripalimab — Toripalimab 240mg ivdrip, every 3 weeks for 6 cycles, with 3 cycles combined with induction chemotherapy, 3 cycles combined with concurrent chemoradiotherapy
  Other Names: JS001
  Arms: Toripalimab+induction chemotherapy +CCRT
Drug: Albumin-bound Paclitaxel — Albumin-bound Paclitaxel 260 mg/m2, d1 of every cycle, every 3 weeks for 3 cycles before radiotherapy
Drug: Cisplatin — Induction cisplatin 80mg/m2, every 3 weeks for 3 cycles before radiotherapy Concurrent cisplatin 100mg/m2, every 3 weeks for 2 cycles during radiotherapy
  Other Names: DDP
Radiation: intensity-modulated radiotherapy — Definitive IMRT of ≥66 Gy will be given .
  Other Names: IMRT

SUMMARY:
This is an open-label, parallel controlled, phase IIa exploratory study that evaluates the efficacy and safety of Toripalimab (PD-1 Antibody) combined with induction chemotherapy （Albumin-bound paclitaxel and cisplatin ）and concurrent chemoradiotherapy in the treatment of nasopharyngeal carcinoma and explores the biomarkers that can predict the efficacy and toxicity of the treatment.

ELIGIBILITY:
Inclusion Criteria:

* Only the patients meeting all the following criteria can be eligible to participate in the trial:

  1. Fully understand this study and voluntarily sign the informed consent form (ICF); have good compliance;
  2. Patients with newly histologically confirmed non-keratinizing nasopharyngeal carcinoma, including WHO II or III ;
  3. locoregionally advanced nasopharyngeal carcinoma (LANPC)（T3-4N0-1M0/T1-4N2-3M0）;
  4. Age 18 to 70 years;
  5. ECOG PS 0-1;
  6. The laboratory examination results before enrollment must meet the following standards:

     1. Neutrophils ≥1.5 × 109 / L;
     2. Platelets ≥100 × 109 / L;
     3. Hemoglobin ≥90g / L (no infusion of concentrated red blood cells within 4 weeks);
     4. Serum creatinine ≤ 1.5 × ULN and creatinine clearance ≥ 60 mL / min;
     5. Total serum bilirubin ≤ 1.5 × ULN;
     6. AST and ALT ≤ 2.5 × ULN;
     7. The ULN of coagulation parameters APTT is not extended for more than 10 seconds, and the ULN of PT is not extended for more than 3 seconds;
  7. Women of childbearing age must confirm that the serum pregnancy test is negative and agree to use effective contraception during drug use and within 1 year after the last dose；Men whose female partners have the ability to become pregnant must agree to use reliable contraception within 1 year from the screening visit to the last Toripalimab administration.

Exclusion Criteria:

1. Women of child-bearing potential are pregnant or breastfeeding ;
2. Have known allergy to large molecule protein products or any compound of Toripalimab;
3. Central nervous system metastases with clinical symptoms accompanied by cerebral edema, requiring hormone intervention, or progression of brain metastases;
4. Prior malignancy within 5 years, except carcinoma in situ of the cervix, adequately treated basal cell carcinoma of the skin and papillary thyroid carcinoma;
5. Received any of the following treatments:

   1. Patients who have been treated with inhibitors of immune regulation (CTLA-4, PD-1, PD-L1, etc.);
   2. Received any research drug within 4 weeks before the first administration of the drug;
   3. Join another clinical study at the same time, unless it is an observational (non-interventional) study or intervention study during follow-up;
   4. Within 28 days before signing the informed consent, received an equivalent dose of >10 mg prednisone/day or other immunosuppressive therapy, and a systemic hormone dose of ≤10 mg prednisone/day or inhaled/topical corticosteroids;
   5. Have been vaccinated with anti-tumor vaccines or have been vaccinated with live vaccines within 4 weeks before the first administration of study drugs;
   6. Have undergone major surgery or severe trauma within 4 weeks before the first administration of study drugs;
6. Uncontrolled clinical symptoms or diseases of the heart, such as: (1) Heart failure above NYHA level II (2) Unstable angina (3) Myocardial infarction occurred within 1 year (4) Clinically supraventricular or Patients with ventricular arrhythmias requiring clinical intervention;
7. Serious infections (CTCAE>2) within 4 weeks before the first use of the study drug, such as severe pneumonia, bacteremia, and infection comorbidities that require hospitalization; baseline chest imaging examinations suggest active lung inflammation . The symptoms and signs of infection exist within 2 weeks before the first dose or require oral or intravenous antibiotic use (excluding prophylactic antibiotic use);
8. Have a history of interstitial lung disease and non-infectious pneumonia;
9. Have active tuberculosis infection, or have a history of active tuberculosis infection within 1 year before enrollment, or have active tuberculosis infection one year ago but have not been formally treated;
10. Have active autoimmune diseases or a history of autoimmune diseases (such as interstitial pneumonia, colitis, hepatitis, pituitary inflammation, vasculitis, nephritis, hyperthyroidism, hypothyroidism, including but not limited to These diseases and syndromes); Autoimmune-mediated hypothyroidism treated with stable doses of thyroid replacement hormone; Type I diabetes with stabilized doses of insulin; but excluding vitiligo or cured childhood asthma/allergy who do not require any intervention in adults;
11. A history of HIV infection, or other acquired, congenital immunodeficiency diseases, or a history of organ transplantation and bone marrow transplantation;
12. Have active hepatitis HBsAg positive and HBV DNA ≥2000IU/ml or 1000 copies/ml, hepatitis C (hepatitis C antibody positive, and HCV-RNA is higher than the detection limit);
13. Known history of psychotropic substance abuse, alcoholism and drug abuse;
14. Any other disease or condition of clinical significance that the investigator believes may affect protocol compliance, or affect the signing of an ICF, or is not suitable for participation in this clinical trial.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-07-15 (Estimated); Primary Completion 2023-12-15 (Estimated); Study Completion 2024-12-15 (Estimated)

PRIMARY OUTCOMES:
Adverse events | 2 years
  Incidence of adverse events as assessed by CTCAE v5.0

SECONDARY OUTCOMES:
Overall survival (OS) | 3 years
  calculated from randomization to the date of death from any cause.
Distant failure-free survival (DFFS) | 3 years
  calculated from randomization to the date of first distant metastasis.
Locoregional failure-free survival (LRFFS) | 3 years
  calculated from randomization to the date of locoregional persistence or 1st locoregional recurrence
Overall response rate （ORR）and Complete response rate（CR） | 2 years
  Defined as percentage of participants achieving complete response (CR) and partial response (PR) according to the RECIST 1.1.
Quality of life (QoL) | 3 years
  The change of QoL from randomization to 12 months after chemoradiation. The European Organization for Research and Treatment of Cancer quality of life questionnaire-C30 (EORTC QLQ-C30）version 3.0 will be used. This questionnaire comprises 30 questions, 24 of which are aggregated into nine multi-question scales, that is, five functioning scales (e.g., physical), three symptom scales (e.g., fatigue) and one global health status scale. The remaining six single-question (e.g., dyspnoea) scales assess symptoms. These 15 scales will be scored according to the official Scoring Manual: 1. Estimate the average of the questions that contribute to the scale; this is the raw score. 2. Use a linear transformation to standardise the raw score, so that scores range from 0 to 100. Thus, a high score for a functional scale represents a high level of functioning, a high score for the global health status represents a high QoL, but a high score for a symptom scale represents a high level of problems.

IPD SHARING:
Plan to Share IPD: No